CLINICAL TRIAL: NCT04207632
Title: Quantifying Muscle Tone in Patients With Brain Injury - a Feasibility Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Elsass Foundation (Other); Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Derek Curtis, Post doctoral fellow, Rigshospitalet, Denmark
Other Study IDs: MMTF123
Record Dates: First submitted 2019-12-19; First posted 2019-12-23 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Treatment Outcome; Muscle Dystonia; Spasticity, Muscle; Muscle Tightness; Acquired Brain Injury; Muscle Tone Abnormalities
Keywords: Shear wave elastography; Portable spasticity assessment device; Feasibility; Outcome measure; Reliability; Validity; Clinimetrics
MeSH Terms: conditions — Dystonia; Muscle Spasticity; Brain Injuries | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intervention: The Group of patients will receive routine treatment of muscle hypertonia with botulinum toxin type A in their elbow flexors.
  Interventions: Drug: Botulinum toxin type A injection

INTERVENTIONS:
Drug: Botulinum toxin type A injection — Ultrasound-guided BoNT-A injection in biceps brachii or brachialis

SUMMARY:
This project will determine the feasibility and validity of measuring elbow muscle flexor stiffness in a population of patients with sub-acute severe acquired brain injury using two measurement methods, the portable spasticity assessment device (PSAD) (Movotec, Charlottenlund, Denmark) and an ultrasound measurement called shear wave sonoelastography (SWE).

DETAILED DESCRIPTION:
The purpose of this study is to investigate the feasibility and validity of measuring hypertonia in the elbow flexors of patients with severe acquired brain injury in their sub-acute rehabilitation and collect data to determine the necessary size for a definitive study to determine the clinimetrics of the test methods. The long-term goal is to establish a valid and clinically feasible method for physiotherapists to quantify muscle tone in patients with neurological disorders.

The study hypotheses are:

1. SWE, PSAD and Modified Ashworth Scale (MAS) measurements can be obtained for elbow flexion hypertonia in all patients (no missing data due to test procedure),
2. SWE and PSAD have a moderate to good intra-day intra-tester reliability (ICC two-way mixed effects model with absolute agreement. ICC>0.5, Bland Altman)
3. Passive muscle stiffness measured using the PSAD and SWE have a fair concurrent validity with MAS (Spearmans correlation >0.3)
4. SWE and PSAD are responsive in measuring a reduction of the effect of routine clinical treatment of the hypertonic muscles with botulinum toxin type A (BTX-A) (paired T-test or Wilcoxon test, p>0.05)

ELIGIBILITY:
The project will include five patients admitted to the clinic for highly specialised neurorehabilitation/TBI. Inclusion criteria for the patients are that they:

1. Fulfil the normal clinical requirements for treatment with BTX-A in at least one of their elbow flexors, (have increased stiffness in at least one of their elbow flexors, MAS greater than 0),
2. Have given the normal informed consent to routine clinical treatment with BTX-A,
3. Have given written informed consent or that proxy consent has been obtained, to participate in the study

Exclusion criteria for patients are that they:

1. Are unable to cooperate with the measurements due to uncontrolled non-voluntary movements
2. Cannot be positioned safely or comfortably for the measurements.

Ages: 5 Years to 99 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients hospitalised for intensive rehabilitation following severe traumatic brain injury with hypertonia in their elbow flexors requirng routine treatment with BoNT-A injection.
Sampling Method: Probability Sample
Enrollment: 5 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2021-01-15 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in resistance to elbow extension measured using the portable spasticity assessment device (PSAD) | Twice at baseline and 4 weeks post BoNT-A injection
  The patient will be measured bilaterally using a PSAD.The PSAD utilises a load cell, gyroscopes and accelerometers and electromyography (EMG) and can measure full passive joint torque and joint angle together with corresponding muscle activity. A reduced passive moment in Nm when moving the joint indicates a reduced tissue stiffness.
Change in muscle stiffness in the treated muscle(s) measured using the shear wave elastography (SWE) | Twice at baseline and 4 weeks post BoNT-A injection
  The patient will be scanned using an ultrasound scanner with shear wave elastography in the treated muscle and the contralateral equivalent. A reduced speed of propgation of the shear waves in m per second indicates a reduced stiffness/tone in the muscle.

SECONDARY OUTCOMES:
Muscle tone measured using modified ashworth scale | Baseline and 4 weeks post BoNT-A injection
  Following standard clinical tone assessment procedure. The scale is from 0 to 4, where a lower value is indicative of a more normal muscle tone.
Passive range of motion | Baseline and 4 weeks post BoNT-A injection
  Passive range of motion in flexion and extension of the elbow joint will be measured. A normal range of motion is associated with normal muscle tone. A reduced range of motion can indicate increased muscle tone.

CONTACTS AND LOCATIONS:
Overall Officials: Derek J Curtis, phd, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to European data regulations